CLINICAL TRIAL: NCT05067946
Title: A Phase 2/3, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of GX-19N, A DNA Vaccine, in Healthy Individuals Who Have Received One of the COVID-19 Vaccines
Brief Title: Evaluation of Efficacy, Safety and Immunogenicity of GX-19N in Healthy Individuals Who Have Received COVID-19 Vaccines
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change of development strategy in consideration of the global COVID-19 situation
Sponsor: Genexine, Inc. (Industry)
Collaborators: PT Kalbe Farma Tbk (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GX-19N-HV-004
Record Dates: First submitted 2021-10-04; First posted 2021-10-05 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — GX-19N vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-19N (Experimental): GX-19N will be intramusculary administered via EP on day 1 and day 29.
  Interventions: Biological: GX-19N
- Placebo (Placebo Comparator): Placebo will be intramusculary administered via EP on day 1 and day 29
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GX-19N — DNA vaccine expressing SARS-CoV-2 S-protein antigen including the Nucleocapsid protein (NP) antigen
  Arms: GX-19N
Other: Placebo — GX-19N formulation buffer
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and immunogenicity of GX-19N in healthy individuals who have received one of COVID-19 vaccine authorized for emergency use.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged 18 years and above at the time of consent
2. Healthy subjects in normal medical condition as determined by medical history, physical examination, and investigator's discretion
3. Have previously received homologous full-dose of COVID-19 vaccine authorized for emergency use, and at least 3 months post second vaccination prior to Day 1
4. Negative results for SARS-COV-2 rapid antigen test at the screening period
5. Able to comply with all study procedures and requirements
6. Agree for blood and nasal swab samples could be collected throughout the study period, including surveillance visit

Exclusion Criteria:

1. Unable to follow clinical and follow-up procedures
2. Acute fever with temperature above 38℃, coughing, breathing difficulty, chills, muscle ache, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to the vaccination
3. History of SARS-CoV-2 infection or have experienced prior administration of an investigational coronavirus (SARS-CoV, MERS-CoV) vaccine
4. History of a malignant disease within the past 5 years
5. Immune dysfunction, including immunodeficiency disorder, or family history of such conditions (Except stable/well-controlled HIV-positive participants)
6. Have received immunoglobulin or blood-derived products within 3 months prior to the vaccination or are scheduled to receive them during the study period
7. Have been dependent on antipsychotic drugs and narcotic analgesics within 6 months prior to the vaccination
8. History or are suspected of alcohol or drug dependency
9. History of hypersensitivity or allergic reactions including anaphylaxis
10. A current or history of clinically significant chronic cardiovascular, endocrine, gastrointestinal, hepatic (including hepatitis B and C), renal, neurological, respiratory, psychiatric or other medical disorders not excluded by other exclusion criteria, that are assessed by the investigator
11. Hemophiliacs or people using anticoagulants who are at a risk of serious bleeding from IM injection
12. Have received or plans to receive other vaccination(s) within 28 days prior to or during study duration (except for influenza vaccine which is not allowed within 14 days before, or 4 weeks after final dose of IP)
13. Have taken an immunosuppressant or immune-modifying drug within 3 months prior to the vaccination; chronic administration (defined as more than 14 continuous days) of immunosuppressant medication within the past 3 months, except topical steroids or short-term oral steroids (course lasting ≤ 14 days)
14. Female who are pregnant or breastfeeding; however, participation is possible if breastfeeding is discontinued prior to participation in the study
15. Have received or have plans to receive other investigational drug(s) while participating in another clinical study or bioequivalence study within 28 days prior to vaccination
16. Not consent to the use of effective contraception at least 90 days after the last vaccination
17. Lack of acceptable sites available for IM injection and EP
18. Deemed ineligible by the investigator based on other clinically significant medical or psychiatric findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
First occurrence of COVID-19 at least 14 days after the second vaccination | Up to 1 year after first vaccination
  Symptomatic, virologically confirmed COVID-19 as described in the study
Incidence of severe solicited adverse events (AEs) | Up to 7 days after each vaccination
  Percentage of subjects reporting grade 3 or higher AEs after each vaccination
Incidence of AEs and Serious AEs (SAEs) after each vaccination | Up to 1 month after each vaccination
  Percentage of subjects reporting AEs and SAEs after each vaccination
Incidence of SAE, and Adverse events of special interest (AESIs), which relevant to COVID-19 including possible vaccine-enhanced disease | Up to 1 year after first vaccination
  SAE and AESIs reported in all subjects at any time after the first vaccination

SECONDARY OUTCOMES:
First occurrence of severe COVID-19 at least 14 days after the second vaccination | Up to 1 year after first vaccination
  Symptomatic, virologically confirmed severe COVID-19 as described in the study
Cell-mediated immune responses after vaccination | Up to 1 year after first vaccination
  Antigen-specific T cell response in a subset of Phase 2/3
Antibody responses after vaccination | Up to 1 year after first vaccination
  Analysis of binding antibodies and neutralizing antibodies in a subset of Phase 2/3

OTHER OUTCOMES:
First occurrence of COVID-19 at least 14 days after the first vaccination | Up to 1 year after first vaccination
  Symptomatic, virologically confirmed COVID-19 as described in the study
First occurrence of asymptomatic, virologically confirmed COVID-19 at least 14 days after the last vaccination in subjects | Up to 1 year after first vaccination
  Without symptom, but virologically confirmed COVID-19 as described in the study

CONTACTS AND LOCATIONS:
Overall Officials: JungWon Woo, Ph.D., Study Director — Genexine, Inc.